CLINICAL TRIAL: NCT03487354
Title: Medical Abortion With Multiple vs Single Daily Dose of Misoprostol in First Trimester Miscarriage: A Randomized Clinical Trial.
Brief Title: Medical Abortion With Single Daily Dose of Misoprostol
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS1753
Record Dates: First submitted 2018-03-25; First posted 2018-04-04 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single daily dose (Active Comparator)
  Interventions: Drug: Misoprostol
- Multiple daily doses (Active Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Misoprostol

SUMMARY:
Medical abortion using multiple vs single daily dose of misoprostol in first trimester miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age more than 18 years old (age of legal consent).
* Gestational age less than 13 weeks.
* Hemoglobin >10 g/dL.
* BMI between 25 kg/m2 and 35 kg/m2.
* Missed abortion.
* Living fetus with multiple congenital malformations incompatible with life.

Exclusion Criteria:

* Maternal age less than 18 years old.
* Gestational age more than 12 weeks.
* Hemoglobin <10 g/dL.
* Anencephaly.
* Fibroid uterus.
* BMI less than 25kg/m2 and more than 35kg/m2.
* Coagulopathy.
* History or evidence of adrenal pathology.
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Complete miscarriage | one week
  Assessed by trans-vaginal ultrasound where endometrial thickness less than 15 mm is considered complete miscarriage

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt